CLINICAL TRIAL: NCT03186183
Title: GPS: Adaptation Trial of an HIV Prevention Counselling Program for HIV-positive and HIV-negative Gay and Bisexual Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Health Initiative for Men (Unknown); Regional HIV/AIDS Connection (Unknown); AIDS Committee of Toronto (Other); Gay ZONE (Unknown); The Ottawa Hospital (Other); University of Victoria (Other); University of Windsor (Other); Ottawa Hospital Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); MAX Ottawa (Unknown)
Responsible Party: Principal Investigator, Trevor Hart, Principal Investigator, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 2016-282
Record Dates: First submitted 2017-05-25; First posted 2017-06-14 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: HIV/AIDS; Sexually Transmitted Infection; Health Behavior
Keywords: HIV prevention; Sexual health; Motivational interviewing; Information-Motivation-Behavioural skills model; Health promotion
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPS program (Experimental): The individual GPS motivational interviewing counseling program has 4-6 sessions.
  Week 1: information on sexually transmitted infections and HIV disclosure laws is reviewed. Participants are introduced to the sex diary, stress exercise, and stages of change model.
  Week 2: a decisional balance exercise about the participant's current sexual behavior is completed and a behavioral goal is chosen.
  Week 3: participants explore their greatest fears and hopes about the goal, and the importance of and their confidence in achieving it.
  Week 4: the facilitator and participant identify triggers, automatic thoughts, counters, strategies, supports, and rewards pertaining to the pursuit of the goal and role play the new goal.
  1-2 supplemental sessions may be added as needed.
  Interventions: Behavioral: GPS program

INTERVENTIONS:
Behavioral: GPS program — GPS is a sexual health promotion and HIV prevention program. It has 4 components: provision of information on HIV and sexually transmitted infections, motivational interviewing counselling, sexual health behavioural skills building, and linkage to care in the local community (e.g., referrals to medical, social service, social, mental health, and substance use programs). Among HIV-positive men who have sex with men (MSM) GPS is associated with positive health outcomes including decreased likelihood of condomless anal sex (CAS), particularly CAS with serodiscordant partners. GPS is also associated with decreased fear of being rejected for insisting on condom use and increased condom use self-efficacy.

SUMMARY:
GPS is a sexual health promotion and HIV prevention peer-delivered counselling program. The GPS program has 4 parts: information provision about HIV and sexually transmitted infections, motivational interviewing counselling, sexual health behavioural skills building, and linkage to care. The adaptation grant has three goals: 1) to establish a multi-region and multi-sectoral team that can deliver the revised program across a variety of settings, 2) to learn how best to deliver this program as individual counselling program and also how to adapt this program for HIV-negative MSM, and 3) to pilot the individual program in 5 settings across Ontario and British Columbia. The research team will evaluate the pilot adaptation through mixed methods, employing a quantitative questionnaire and one-on-one semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* self-identify as a man
* self-identify as gay, bisexual, queer, same-gender-loving, or a man who has sex with men
* report having engaged in condomless anal sex in the last 3 months
* able to speak, read, and aurally comprehend English
* depending on the study site, report HIV-negative or HIV-positive status

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as a man; transmen are welcome
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change in the number of serodiscordant condomless anal sex acts | Past 2 months (measured at baseline, post-treatment, and 3-month follow-up)
  Participants will be asked to report the number of times they engaged in anal sex in the without a condom with a partner of opposite or unknown HIV status in the past two months as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.

SECONDARY OUTCOMES:
Change in the number of sexual partners | Past 2 months (measured at baseline, post-treatment, and 3-month follow-up)
  Participants will be asked to report the number of sexual partners they had who are HIV-positive, HIV-negative, and of unknown HIV status in the past two months as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.
Change in the number of receptive condomless anal sex acts | Past 2 months (measured at baseline, post-treatment, and 3-month follow-up)
  Participants will be asked to report the number of times they engaged in receptive anal sex without a condom in the past two months as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.
Change in the number of insertive condomless anal sex acts | Past 2 months (measured at baseline, post-treatment, and 3-month follow-up)
  Participants will be asked to report the number of times they engaged in insertive anal sex without a condom in the past two months as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.
Change in HIV viral load status | Most recent viral load test (asked at baseline, post-treatment, and 3-month follow-up)
  HIV-positive participants will be asked to report whether they had a detectable or undetectable HIV viral load at their last viral load test as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.
Change in use of HIV pre-exposure prophylaxis (PrEP) | Present use (asked at baseline, post-treatment, and 3-month follow-up)
  For HIV-negative participants, participants will be asked whether they use HIV PrEP as part of a self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.

OTHER OUTCOMES:
Change in loneliness | Present loneliness (measured at baseline, post-treatment, and 3-month follow-up)
  Measured using the University of California, Los Angeles Loneliness Scale, which is part of the self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.
Change in sexual compulsivity | Present sexual compulsivity (measured at baseline, post-treatment, and 3-month follow-up)
  Measured using the Sexual Compulsivity Scale, which is part of the self-report questionnaire. This self-report questionnaire is administered at baseline, post-treatment (which is approximately 6 weeks after baseline), and at 3-month follow-up in order to measure changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Hart, PhD, Principal Investigator — Toronto Metropolitan University
Locations (6):
- Canada (6):
  - Health Initiative for Men, Vancouver, British Columbia
  - Regional HIV/AIDS Connection, London, Ontario
  - Immunodeficiency Clinic - The Ottawa Hospital, Ottawa, Ontario
  - Gay ZONE (Centretown Community Health Centre), Ottawa, Ontario
  - MAX Ottawa, Ottawa, Ontario
  - AIDS Committee of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No